CLINICAL TRIAL: NCT02770859
Title: Per-Oral Endoscopic Myotomy (POEM) for the Treatment of Achalasia, Database Repository
Acronym: POEM
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John DeWitt, Director, Endoscopic Ultrasound, Indiana University
Other Study IDs: 1410540149
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Achalasia
Keywords: Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — nephronectin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: POEM (Per Oral Endoscopic Myotomy) — Per-Oral endoscopic myotomy (creating a muscle [esophagus] opening), an incision-less (no cutting of the surface of the body) endoscopic procedure, is an effective non-surgical alternative to release the muscle & sphincter of the LES for the treatment of achalasia
  Other Names: POEM

SUMMARY:
POEM (Per-Oral endoscopic myotomy (creating a muscle [esophagus] opening), an incision-less (no cutting of the surface of the body) endoscopic procedure, is an effective non-surgical alternative to release the muscle & sphincter of the LES for the treatment of achalasia.

DETAILED DESCRIPTION:
Achalasia is a disease of the muscle of the esophagus (food tube) & means "a failure to relax." The esophagus consists of 3 parts: the first part (uppermost part) is the upper esophageal sphincter (UES). The UES is a specialized ring of muscle which separates the esophagus from the throat, & prevents food in the second part (body) of the esophagus from regurgitating into the throat. The third part of the esophagus (lower esophageal sphincter [LES]) also consists of a specialized ring of muscle which separates the body of the esophagus from the stomach, & prevents food & acid from regurgitating into the body of the esophagus. When achalasia is present, patients experience dysphasia (difficulty swallowing food, & [sometimes] liquids), chest pain & can experience recurrent pneumonia & loss of weight.

Current treatments for achalasia include oral medications (calcium channel blockers) to relax the LES (difficult to swallow pill/capsule), dilation (stretching) of the LES, (temporary relief) & Esophagomyotomy (general surgery to cut the LES).

POEM (Per-Oral endoscopic myotomy (creating a muscle [esophagus] opening), an incision-less (no cutting of the surface of the body) endoscopic procedure, is an effective non-surgical alternative to release the muscle & sphincter of the LES for the treatment of achalasia.

ELIGIBILITY:
Inclusion Criteria:

18 years of age Referral for the treatment of Achalasia

Exclusion Criteria:

Less than 18 years of age; Absence of Achalasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 with demonstrated symptoms of Type II or Type III achalasia.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-10-16 (Actual); Primary Completion 2040-01-31 (Estimated); Study Completion 2040-01-31 (Estimated)

PRIMARY OUTCOMES:
Improved Eckardt Score | 5 years
  Consists of 4 questions used to characterize the severity of achalasia. The questions include symptoms related to dysphagia, chest pain, regurgitation, and weight loss. Each question is assigned a score from 0 to 3 based on the patient's self reported response.
  The overall score ranges from 0-12, with anything less than 3 meaning no active symptoms, and anything higher than a 3 suggestive of active symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: John M DeWitt, M.D., Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] DeWitt J, Stainko S, Perkins A, Rosenheck M, Al-Haddad M. Impact of prior endoscopic or surgical interventions on clinical outcomes after peroral endoscopic myotomy for achalasia. Surg Endosc. 2026 Jan;40(1):174-181. doi: 10.1007/s00464-025-12258-3. Epub 2025 Oct 6. PMID 41051511
- [Derived] Jacobs CC, Al-Haddad M, Stainko S, Perkins A, DeWitt JM. Prevalence and impact of opioid use in patients undergoing peroral endoscopic myotomy. Gastrointest Endosc. 2023 Apr;97(4):655-663.e2. doi: 10.1016/j.gie.2022.12.006. Epub 2022 Dec 9. PMID 36509112
- [Derived] DeWitt JM, Kessler WR, Wo JM, Stainko S, Perkins A, Dickason D, Al-Haddad MA, Siwiec R. Symptom Association for Gastroesophageal Reflux Disease by pH Monitoring After Peroral Endoscopic Myotomy. Am J Gastroenterol. 2022 Aug 1;117(8):1316-1319. doi: 10.14309/ajg.0000000000001801. Epub 2022 Apr 25. PMID 35467562
- [Derived] DeWitt JM, Siwiec R, Kessler WR, Wo JM, Stainko S, Picklesimer Doyle M, Perkins A, Dickason D, Al-Haddad MA. Comparison of functional lumen imaging probe and high-resolution manometry to assess response after peroral endoscopic myotomy. Gastrointest Endosc. 2022 May;95(5):855-863. doi: 10.1016/j.gie.2021.12.029. Epub 2022 Jan 1. PMID 34979118